CLINICAL TRIAL: NCT00103350
Title: A Phase 1-2, Multicenter, Randomized, Double-Blind, Placebo Controlled, Prospective Study to Evaluate the Safety and Potential Efficacy of Single, Increasing Doses of TG100-115 in Subjects Undergoing Percutaneous Coronary Intervention for Acute Anterior ST Elevation Myocardial Infarction
Brief Title: Safety of TG100-115 for Heart Attack Treated With Angioplasty
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TargeGen (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TG001-03; NCT00104208 (obsolete NCT alias)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; infarct size; angioplasty; percutaneous coronary intervention; Acute Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — 3-(2,4-diamino-6-(3-hydroxyphenyl)pteridin-7-yl)phenol

INTERVENTIONS:
Drug: TG100-115

SUMMARY:
TG100-115 is able to reduce the size of heart attacks in pre-clinical models. The hypothesis of this study is that TG100-115 can be given safely to patients who suffer a heart attack and undergo angioplasty to restore blood flow. We will also evaluate whether TG100-115 reduces heart muscle damage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 yrs
* ECG patterns consistent with an acute anterior myocardial infarction with ST segment elevation of 2mm in two contiguous ECG leads among leads V1-V4.
* Have prolonged, continuous (lasting at least 20 mins) signs and symptoms of myocardial ischemia not eliminated with nitrates.
* Intent to proceed to primary PCI within 6 hours of chest pain onset
* Sign an informed consent form and be willing to attend follow-up visits for safety and other study assessments.

Exclusion Criteria:

* Female of childbearing potential.
* History of previous myocardial infarction.
* History of congestive heart failure.
* Requirement for a cardiac pacemaker or defibrillator.
* Cardiogenic shock.
* Patients previously treated with thrombolytic therapy.
* Myocardial ischemia precipitated by a condition other than atherosclerotic coronary artery disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Safety and pharmacokinetics of TG100-115

SECONDARY OUTCOMES:
Impact of TG100-115 on infarct size

CONTACTS AND LOCATIONS:
Locations (1):
- David Holmes, MD, Rochester, Minnesota, United States